CLINICAL TRIAL: NCT05559567
Title: Axial Length With Adult Onset Myopia
Brief Title: Axial Length With Adult Onset Myopia (ALWAOM)
Acronym: ALWAOM
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Art Optical Contact Lens, Inc. (Industry)
Collaborators: University of Missouri, St. Louis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ALWAOM2022
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Myopia
Keywords: Axial Length; Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Orthokeratology (Other): Orthokeratology is fitting of a contact lens for overnight wear to flatten the cornea and correct myopia temporarily during the day. This procedure has also been shown to slow down the axial length growth in children.
  Interventions: Device: Orthokeratology

INTERVENTIONS:
Device: Orthokeratology — The use of a specialty GP contact lens to temporarily correct myopia

SUMMARY:
Purpose: To determine axial length progression and its relationship with myopia onset and progression in adults.

DETAILED DESCRIPTION:
Objectives

1. Determine axial length progression over a two year period of at least 100 subjects/students aged 21 or over (subjects may come from multiple sites). Subjects are to be chosen from optometric education programs beginning in the student's first year.
2. Determine correlation of axial length changes to refractive changes over the two year period.
3. Obtain results of orthokeratology and its effect on axial length and refractive changes.

Methods

1. Measurements of axial length with optical biometry will be taken at yearly intervals for three years and recorded on a spreadsheet (see attached) for future data analysis. Effort will be made to perform measurements at approximately same date each year.
2. Refractive error will be measured using a consistent method such as an autorefractor at yearly intervals for three years and recorded on same spreadsheet as axial length for future data analysis. Effort will be made to perform measurements at approximately same date each year.
3. Subjects that are fit into orthokeratology will be fit with the MOONLENS design (provided by Art Optical at no charge) per normal fitting protocol and followed up with normal protocol Axial length will be measured pre-fitting and at least every year for the three year period. Topography will be captured at pre-fitting and post fitting per normal protocol with images taken at least once per year for three year period. Refraction will also be conducted at least once per year. Axial length and refraction data are to be recorded on same spreadsheet as above and topography saved to a separate folder for future analysis.

ELIGIBILITY:
Inclusion Criteria:

1. 1st year optometry student
2. Refractive error - spherical Component: +2.00D to -5.00D; astigmatic Component: up to -1.50D; non-presbyopic
3. Not currently using any treatment for myopia control, including Orthokeratology lenses, soft multifocal lenses, MiSight lenses, pharmacological interventions, or spectacles for myopia control
4. No significant anterior or posterior segment disease

Exclusion Criteria:

1. Non-graduate student
2. Refractive error outside of: +2.00D to -5.00D; astigmatic Component: up to -1.50D; presbyopic
3. Any participants using treatment for myopia control, including Orthokeratology lenses, soft multifocal lenses, MiSight lenses, pharmacological interventions, or spectacles for myopia control
4. Significant anterior or posterior segment disease
5. Pregnancy
6. Significant systemic disease that may affect refractive error (i.e. diabetes)

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Axial Length progression | Two years
  The change in the length of the eye from the anterior cornea to the retina over time
Effect of Orthokeratology on axial length changes | Two years
  Compare the average axial length changes of subjects wearing orthokeratology lenses to those who do not

CONTACTS AND LOCATIONS:
Locations (1):
- University of Missouri-St. Louis College of Optometry, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No